CLINICAL TRIAL: NCT03473262
Title: Efficacy and Safety of Empagliflozin vs. Insulin Glargine add-on Therapy in Patients With Inadequately Controlled Type 2 Diabetes Under Triple Combination Therapy
Brief Title: Empagliflozin-based Quadruple Combination vs Insulin Glarine-based Combination Therapy in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Chungbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Eu Jeong Ku, ChungbukNUH, Chungbuk National University Hospital
Other Study IDs: 2017-03-011; eujeongku (Registry Identifier: Eu Jeong Ku)
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; Sodium glucose cotransporter 2 inhibitor; Empagliflozin; Insulin glargine
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EMPA: Empagliflozin 25 mg/day
- INS: Insulin Glargine dose-titrated

SUMMARY:
This study evaluates the efficacy and safety of the empagliflozin as add-on thearpy compared to insulin glargine-based antidiabetic agents (OADs) combination thearpy in patients with type 2 diabetes inadequately controlled on triple OADs in a real clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Are inadequately controlled with triple OADs (metformin, sulfonylurea, dipeptidyl peptidase inhibitor) as evidenced by HbA1c >7.5% and <12.0%

Exclusion Criteria:

* Type 1 diabetes
* Gestional diabetes
* Diabetes due to secondary causes
* Receiving anticancer treatment
* Receiving glucocorticoids or immune-suppressants
* Have been treated with sodium glucose co-transporter 2 inhibitors for more than 7 consecutive days within 3 months before entering the study
* Have been treated with any type of insulin for more than 7 consecutive days within 3 months before entering the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targeted population consists of adult patients with type 2 diabetes mellitus treated in outpatient setting by specialists.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c From Baseline to Week 24 | Baseline, Week 24
Changes in Fasting Plasma Glucose From Baseline to Week 24 | Baseline, Week 24

SECONDARY OUTCOMES:
Percentage of Patients Who Achieved Glycemic Target of HbA1c ≤7.0% at Week 24 | Baseline, Week 24
Changes in HbA1c From Baseline to Week 12 | Baseline, Week 12
Changes in Fasting Plasma Glucose From Baseline to Week 12 | Baseline, Week 24
Changes in Weight Between Baseline and Week 24 | Baseline, Week 24
Changes in Body Mass Index Between Baseline and Week 24 | Baseline, Week 24
Changes in Total Cholesterol Between Baseline and Week 24 | Baseline, Week 24
Changes in HDL Cholesterol Between Baseline and Week 24 | Baseline, Week 24
Changes in LDL Cholesterol Between Baseline and Week 24 | Baseline, Week 24
Changes in Triglycerides Between Baseline and Week 24 | Baseline, Week 24
Changes in Systolic Blood Pressure Between Baseline and Week 24 | Baseline, Week 24
Changes in Dystolic Blood Pressure Between Baseline and Week 24 | Baseline, Week 24
Percentage of Patients With Hypoglycemia Episodes Between Baseline and Week 24 | Baseline, Week 24
  All episodes consistent with hypoglycemia with or without a confirmatory blood glucose reading were collected.
Percentage of Patients With At Least 1 Episode of Genitourinary Tract Infections Between Baseline and Week 24 | Baseline, Week 24

IPD SHARING:
Plan to Share IPD: No